CLINICAL TRIAL: NCT04357223
Title: A Parallel, Randomised, Double Blind, Placebo Controlled Study to Investigate the Effect of NOGO on Overactive Bladder in Men and Women
Brief Title: NOGO for an Overactive Bladder
Acronym: NOGO-OAB
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: SagaNatura (Industry)
Collaborators: Universidad Politecnica de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Saga-002
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Overactive Bladder; Nocturia
MeSH Terms: conditions — Urinary Bladder, Overactive; Nocturia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental)
  Interventions: Drug: extract from Angelica archangelica leaf
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: extract from Angelica archangelica leaf — A standardized extract from Angelica archangelica leaf. Capsule, Twice Daily
  Arms: Experimental
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized and placebo-controlled study to evaluate the safety and effectiveness of NoGo, a standardized extract from Angelica archangelica, on overactive bladder

ELIGIBILITY:
Inclusion Criteria:

* Suspected or diagnosed with overactive bladder (average ≥ of 1.5 nocturnal voids per night and/or less then 2 hours between voids at least half time of the day (question 2 IPSS)

Exclusion Criteria:

* High alcohol consumption (males > 3 beers/day (36 g alcohol), females >2 beers/day --
* (24 g alcohol), but we take weekly average.
* Abnormal urinary findings suggestive of urinary tract infection, significant hematuria or glucosuria requiring further evaluation.
* Chronic incontinence.
* Recurrent urinary tract infections (3 or more times per year).
* Pregnancy, lactation, last child born at least one year before, uterine prolapse, histerectomy
* Surgical treatment for bladder outlet obstruction/BPH performed within the past 6 months. Moderate to severe prostate hyperplasia (IPSS questionnaire).
* Medical history or active conditions which, in the opinion of the principal investigator (PI) and physicians participating in the study would prohibit participation in the study. This includes, but is not limited to: diabetes, cancer, renal failure, cirrhosis or chronic liver disease, pancreatic diseases, recent (<6 months) myocardial infarction or unstable coronary artery disease.
* Psychiatric diseases and medication.
* Use of NoGO or other products containing A. archangelica extract within the previous 2 months prior to randomisation.
* Known allergy to compound or any other ingredients of NoGo.
* Supplements like pumpkin seeds, natural products with diuretic effect. Not exclusion if they have a wash out period.
* Receipt of an investigational product within 30 days prior to enrolment or expected receipt during this study.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Reduction of urination frequency (number of voids per 24 hours) | 6 weeks
  Reduction in number of voids per 24 hours as assessed by a 3 day voiding diary before and after treatment

SECONDARY OUTCOMES:
Reduced number of daytime voids | 6 weeks
  Reduction in number of voids occurring during waking hours as assessed by a 3 day voiding diary before and after treatment
Reduced number of nocturnal voids (nocturia) | 6 weeks
  Reduction in number of voids occurring during sleeping hours as assessed by a 3 day voiding diary before and after treatment
Reduced number of nocturnal voids (nocturia) per hour sleeping time | 6 weeks
  Reduction in number of voids occurring during sleeping hours corrected by sleeping time as assessed by a 3 day voiding diary before and after treatment
Reduced number of voids occurring shortly after the last one | 6 weeks
  Reduction in number of voids occurring shortly after the preceding void (less than 60, 90 and 120 minutes) as assessed by a 3 day voiding diary before and after treatment
Improvement of the results of the International Consultation on Incontinence Questionnaire Overactive Bladder Module (ICIQ-OAB) | 6 weeks
  Questionnaire assessing overactive bladder. Overall score is 0-16 with greater values indicating increased symptom severity
Improvement of the results of the The International Prostate Symptom Score (IPSS) | 6 weeks
  A questionnaire assessing prostate symptoms. Overall score is 0-35 (7 questions with score 0-5 each), with greater values indicating increased symptom severity

CONTACTS AND LOCATIONS:
Overall Officials: Marcela Gonzalez-Gross, Ph.D., Principal Investigator — INEF- Universidad Politecnica de Madrid
Locations (1):
- Universidad Politecnica de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lopez-Seoane J, Gesteiro E, Castro-Alija MJ, Quesada-Gonzalez C, Perez-Ruiz M, Gonzalez-Gross M. Effects of Angelica archangelica Extract on Overactive Bladder: A Pilot Randomized Controlled Trial. Food Sci Nutr. 2025 Dec 8;13(12):e71258. doi: 10.1002/fsn3.71258. eCollection 2025 Dec. PMID 41368330